CLINICAL TRIAL: NCT05941611
Title: Results of Objective Brushing Data Recorded From a Powered Toothbrush Used by Elderly Individuals With Mild Cognitive Impairment Related to Values for Oral Health
Brief Title: Results From Objective Brushing Data Saved From a Powered Toothbrush Related to Values for Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blekinge Institute of Technology (Other)
Collaborators: Kristianstad University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BTH-6.1.1-0084-2023
Record Dates: First submitted 2023-06-13; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Gingivitis; Periodontal Diseases
Keywords: Mild Cognitive Impairment; Oral Health; Powered toothbrush
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partisipants (Experimental)
  Interventions: Device: Powered toothbrush

INTERVENTIONS:
Device: Powered toothbrush — Oral-B powered toothbrush

SUMMARY:
For this study, 213 individuals were recruited. During the Baseline examination, each participant received a powered toothbrush and was carefully instructed on how to use the toothbrush and recommended using it for at least 2 minutes every morning and evening. No restrictions were imposed on the use of other oral health products. The study lasted from June 2018 to October 2020 and included a screening, a baseline examination, and additional reexaminations at 6 and 12 months. The Oral-B application was installed on the participant's mobile phones or computer tablets. Participants were instructed verbally and in writing on transferring data from the powered toothbrush to the application. The present study aimed to investigate how the true use of the powered toothbrush, in terms of frequency and duration, affects plaque index (PI), bleeding on probing (BOP), and periodontal pocket depth (PPD) ≥4 mm in a group of elderly individuals with MCI. A second aim was to compare the registered time and brush frequencies to the individual's self-estimated usage of the powered toothbrushes.

ELIGIBILITY:
Inclusion Criteria:

* Being 55 years or older
* Having experienced memory problems in the last six months before inclusion
* Having a Mini-Mental State Examination score of 20-28
* Are not receiving any formal care
* Having at least ten teeth of their own

Exclusion Criteria:

* Having a terminal illness with less than three years of expected survival
* Having another known significant cause of disease explaining cognitive impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change in the amount of dental plaque | From Baseline to month 6 and to month12
  Plaque Index in percent
Change in the amount of gingival bleeding on probing | From Baseline to month 6 and to month12
  Number of bleeding from the gingiva measured on four sides of the teeth presented as a percentage
Change in the number of periodontal pockets 4 mm or deeper | From Baseline to month 6 and to month12
  The number of periodontal pockets 4 mm or deeper measured on four of the tooth surfaces presented as a percentage
Change of average brush time | From Baseline to month 6 and to month12
  The average time used for tooth brushing presented in min and sec.
Change in the number of brush sessions | From Baseline to month 6 and to month12
  The number of uses of the toothbrush per day

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sanmartin-Berglund, Professor, Study Chair — Blekinge Institute of Technology
Locations (1):
- Blekinge Institute of Technology, Karlskrona, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analyzed during the current study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Starting after publication
Access Criteria: The datasets used and analyzed during the current study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Flyborg J, Renvert S, Anderberg P, Larsson T, Sanmartin-Berglund J. Results of objective brushing data recorded from a powered toothbrush used by elderly individuals with mild cognitive impairment related to values for oral health. Clin Oral Investig. 2023 Dec 21;28(1):8. doi: 10.1007/s00784-023-05407-2. PMID 38123762